CLINICAL TRIAL: NCT00427505
Title: An Open-label, One-sequence Cross-over Study to Investigate the Effect of Deferasirox on the Pharmacokinetics of Midazolam in Healthy Volunteers
Brief Title: Study to Investigate the Effect of Deferasirox on the Pharmacokinetics of Midazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: e, Novartis Pharmaceuticals
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A2126
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2009-11-19 (Estimated); Status verified 2009-11

CONDITIONS: Healthy
Keywords: Interaction; healthy volunteers; deferasirox; midazolam
MeSH Terms: interventions — Deferasirox

INTERVENTIONS:
Drug: Deferasirox

SUMMARY:
This is a study to investigate the pharmacokinetics of deferasirox

ELIGIBILITY:
Inclusion Criteria:

* Good health
* No evidence of iron deficiency
* Weight between 50 and 100 kg
* Body Mass Index between 19 and 29 kg/m2

Exclusion Criteria:

* Use of certain drugs, herbal remedies or nutrients

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22
Dates: Start 2006-07

PRIMARY OUTCOMES:
To assess the effect of deferasirox on the pharmacokinetics of midazolam

SECONDARY OUTCOMES:
Safety assessed by adverse events (AEs)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis